CLINICAL TRIAL: NCT04136340
Title: Virtual Visits by Supportive Care Specialists to Cancer Patients at Home: A Randomized Controlled Pilot Noninferiority Trial of Video Telemedicine
Brief Title: Supportive Care Delivered by Telemedicine to Cancer Patients at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-382
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Cancer; Supportive Care
Keywords: Telemedicine; Virtual Visits; 19-382
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Noninferiority, randomized, controlled trial (RCT) in which all patients will meet with a supportive care specialist in-person for the initial clinic visit, and then receive follow-up supportive care visits either in-person at clinic or via home video telemedicine.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person follow-up (Active Comparator): Due to the COVID-19 pandemic, patients originally randomized to the in-person group received telemedicine visits. Thus, the researchers will expand our sample for these interviews to include patients who have completed at least 2 telemedicine follow-up visits whether they were originally randomized to the in-person group or the home telemedicine group.
  Interventions: Other: In-person in clinic follow-up visit
- Home Telemedicine follow-up (Experimental)
  Interventions: Other: Telemedicine follow-up visit

INTERVENTIONS:
Other: In-person in clinic follow-up visit — Patient will be seen in-person (i.e. an IR/NV or AFX visit) in the clinic by a Supportive Care Specialist for at least 3 follow-up visits over 14 weeks. Any patients randomized to the in-person group who experience an extraordinary burden and/or are physically unable to attend their in-person visits will be able to be seen by their Supportive Care Service clinician via a home telemedicine visit (patients will return to their original group assignment if possible).
  Arms: In-person follow-up
Other: Telemedicine follow-up visit — i. Patients will be seen by video telemedicine at home by a Supportive Care Specialist for at least 3 follow-up visits over 14 weeks.
  ii. Patients will have access to a clickable link that will initiate a video telemedicine call to the clinician's office. The clinical team will be responsible for answering such calls and for ensuring the clinician and the patient connect and begin the actual visit.
  Arms: Home Telemedicine follow-up

SUMMARY:
This study will test whether supportive care follow-up delivered to cancer patients at home by telemedicine ("virtual" medical visits using telecommunications technologies) is as effective as in-person supportive care visits in the clinic.

DETAILED DESCRIPTION:
The protocol was developed and initially implemented when the standard of care for Supportive Care (and oncology) follow-up at MSK was in-person visiting and home telemedicine was only in an early stage of use at the institution. During the COVID-19 crisis, all outpatient Supportive Care visits and most oncology visits at MSK have been handled via telemedicine to protect patient (and staff) safety.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* solid tumor of any type
* completed an initial in-person clinic visit (i.e. an IR/NV or AFX visit) at Rockefeller Outpatient Pavilion with Dr. Saldivar, Dr. Martin, Supportive Care physicians, or Andrea Dolan, a Supportive Care nurse practitioner
* planned for Supportive Care Service follow-up visits, but none yet completed
* enrolled on the MyMSK secure online patient portal and have access to the portal off site of MSK campuses
* resident of New York or New Jersey or Connecticut (clinicians may not be licensed in other states, as would be required for televisits to patients there)

Exclusion Criteria:

* Patients and informal caregivers who cannot communicate with clinicians/respond to instruments in English without the use of an interpreter

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Health-Related Quality of Life: FACT-G | Week 14
  will be used to quantify health-related quality of life at baseline and Week 14 after randomization. All items in the FACT-G use a 5-point scale (0=Not at all to 4=Very much) and the total score sums four subscales and ranges from 0-108 (higher=better QoL). Change in total score at Week 14 after randomization vs. baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Nelson, MD,JD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm